CLINICAL TRIAL: NCT02164201
Title: Post Market Surveillance Study Evaluating the Operative Management of Anastomotic Bleeding by Means of an Adjunctive Application of BioFoam Surgical Matrix in Cardiovascular Surgery
Brief Title: Post Market Surveillance Study Evaluating BioFoam Surgical Matrix in Cardiovascular Surgery
Status: Completed | Type: Observational
Sponsor: CryoLife Europa (Industry)
Responsible Party: Sponsor
Other Study IDs: BFM1301.000-M
Record Dates: First submitted 2014-06-12; First posted 2014-06-16 (Estimated); Last update posted 2015-07-29 (Estimated); Status verified 2015-07

CONDITIONS: Cardiovascular Procedures; Thoracic Aortic Aneurysm; Aortic Valve Replacement; Type A Aortic Dissection
Keywords: Type A Aortic Dissection (where the use of BioFoam is limited to the anastomotic site)
MeSH Terms: conditions — Aortic Aneurysm, Thoracic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a prospective, multicenter, single-arm study designed to collect clinical data to support the safety and effectiveness of BioFoam used as a surgical adjunct to anastomotic hemostasis following cardiovascular surgery.

The overall objective of this clinical study is to collect clinical data supporting the safety and effectiveness of BioFoam used as a surgical adjunct to anastomotic hemostasis following cardiovascular surgery. This study is intended as a post-market surveillance (follow-up) study.

ELIGIBILITY:
Inclusion Criteria:

* Subject is undergoing an elective cardiac or cardiovascular procedure;
* Subject is willing and able to give prior written informed consent for investigation participation; and
* Subject is > 18 years of age.

Intraoperative inclusion criteria include:

• Subject that requires the use of an adjunctive surgical hemostatic agent to the repair site to control generalized oozing following standard repair procedures (such as sutures and staples).

Exclusion Criteria:

* • Subject with known hypersensitivity to albumin, bovine products, or glutaraldehyde;

  * Subject with active infection (either systemic or in the repair region);
  * Subject whose pathology or underlying disease state makes them an unacceptable candidate for a clinical investigation in the opinion of the Investigator;
  * Subject diagnosed with a coagulation disorder;
  * Subject with abnormal calcium metabolism (e.g., chronic renal failure, hyperparathyroidism);
  * Subject whose life expectancy is less than that required for the prescribed follow-up duration;
  * Subject who is pregnant, planning on becoming pregnant during the follow-up period, or actively breast-feeding; or
  * Subject who is immunocompromised.

Intraoperative exclusion criteria include:

• Any major intraoperative bleeding incidences (i.e., American College of Surgeons Advanced Trauma Life Support Class II, III, or IV Hemorrhage).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing cardiac or cardiovascular procedures, including, but not limited to:
  Thoracic Aortic Aneurysm Aortic Valve Replacement Type A Aortic Dissection (where BioFoam is limited to the anastomotic site)
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2014-08; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Achievement of haemostasis | 3 minutes after application

SECONDARY OUTCOMES:
Time to haemostasis | measured through to 10 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Bernhard Voss, PD Dr Med, Principal Investigator — Deutsches Herzzentrum Muenchen; Ottavio Alfieri, Professor, Principal Investigator — San Raffale Hospital
Locations (2):
- German Heart Center, Munich, Germany
- San Raffale Hospital, Milan, Italy